CLINICAL TRIAL: NCT03781804
Title: A 24-Week Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study Evaluating the Efficacy and Safety of Intranasal Administration of 186 and 372 μg of OPN-375 Twice a Day (BID) in Subjects With Chronic Rhinosinusitis With or Without the Presence of Nasal Polyps
Brief Title: Study Evaluating the Efficacy and Safety of Intranasal Administration of OPN-375 in Subjects With Chronic Rhinosinusitis With or Without the Presence of Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-CS-3205
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPN-375 186 μg BID (Active Comparator): OPN-375 186 μg BID x 24 Weeks
  Interventions: Drug: OPN-375
- OPN-375 372 μg BID (Active Comparator): OPN-375 372 μg BID x 24 Weeks
  Interventions: Drug: OPN-375
- Placebo (Placebo Comparator): Matching Placebo BID x 24 Weeks
  Interventions: Drug: OPN-375

INTERVENTIONS:
Drug: OPN-375 — OPN-375, BID

SUMMARY:
This is a 24-week randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of intranasal administration of 186 and 372 μg twice daily (BID) of OPN-375 in subjects with chronic rhinosinusitis (CS) with or without nasal polyps.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of intranasal administration of twice-daily doses of 186 and 372 µg of OPN-375 (fluticasone propionate) with placebo in subjects with chronic rhinosinusitis using the following co-primary endpoints:

1. A change from baseline in symptoms as measured by a composite score of nasal congestion, facial pain or pressure sensation, and nasal discharge (anterior and/or posterior) at the end of Week 4.
2. A change from baseline to Week 24/Early Termination (ET) in the average percent of the volume opacified in the ethmoid and maxillary sinuses.

ELIGIBILITY:
Potential subjects must meet the following criteria to enter this study:

1. men or women aged 18 years and older at baseline visit
2. women of childbearing potential must be abstinent, or if sexually active,

   1. be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   2. be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   3. be postmenopausal (amenorrhea for at least 1 year)
3. women of child-bearing potential must have a negative urine pregnancy test at Visit 1 (Screening)
4. must have a history of chronic rhinosinusitis (CRS) and be currently experiencing 2 or more of the following symptoms, 1 of which has to be either nasal congestion or nasal discharge (anterior and/or posterior nasal discharge) for equal to or greater than 12 weeks:

   * nasal congestion
   * nasal discharge (anterior and/or posterior nasal discharge)
   * facial pain or pressure
   * reduction or loss of smell
5. endoscopic evidence of nasal mucosal disease, with edema, purulent discharge, or polyps in middle meatus, bilaterally, or presence of bilateral disease on a prior computed tomography (CT) scan performed within 14 days of Visit 1
6. must have confirmatory evidence via a CT scan of bilateral sinus disease (have at least 1 sinus on each side of nose with a Lund-Mackay score of ≥1)
7. baseline CT scan must show a combined ≥25% opacification of the ethmoid sinuses and ≥25% opacification of at least 1 maxillary sinus
8. must have at least moderate symptoms (as defined in protocol) of nasal congestion as reported by the subject, on average, for the 7-day period preceding Visit 1 (Screening) run-in
9. must have an average morning score of at least 1.5 for congestion on the Nasal Symptom Scale (as defined in protocol) recorded on the subject diary over a 7-day period during the first 14 days of the single-blind run-in period
10. must demonstrate an ability to correctly complete the daily diary during the run-in period to be eligible for randomization
11. Subjects with comorbid asthma or chronic obstructive pulmonary disorder (COPD) must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use) within the 3 months before Visit 1 (Screening). Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent) for at least 3 months before Visit 1 (Screening) with plans to continue use throughout the study.
12. Subjects with aspirin-exacerbated respiratory disease, who have undergone aspirin desensitization and are receiving daily aspirin therapy, must be receiving therapy for at least 6 months prior to Visit 1.
13. must be able to cease treatment with intranasal steroids, inhaled corticosteroids (except permitted doses listed above for asthma and COPD) at the screening visit
14. must be able to cease treatment with oral and nasal decongestants and antihistamines at Visit 1 (Screening)
15. must be able to use the exhalation delivery system (EDS) correctly; all subjects will be required to demonstrate correct use with the practice EDS at Visit 1 (Screening).
16. must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Potential subjects who meet any of the following criteria will be excluded from entering this study:

1. women who are pregnant or lactating
2. inability to have each nasal cavity examined for any reason, including nasal septum deviation
3. inability to achieve bilateral nasal airflow
4. is currently taking XHANCE®
5. have previously used XHANCE for more than 1 month and did not achieve an adequate symptomatic response
6. the nasal/sinus anatomy prevents the accurate assessment of sinus volume via CT scan
7. history of sinus or nasal surgery within 6 months before Visit 1 or has not healed from a prior sinus or nasal surgery
8. have current evidence of odontogenic sinusitis, sinus mucocele (the affected sinus is completely opacified and either the margins are expanded and/or thinned OR there are areas of complete bone resorption resulting in bony defect and extension of the "mass" into adjacent tissues), evidence of allergic fungal sinusitis, or evidence of complicated sinus disease (including, but not limited to, extension of inflammation outside of the sinuses and nasal cavity)
9. have a paranasal sinus or nasal tumor
10. have a polyp extending outside the ostiomeatal complex/middle turbinate (anterior or inferior) that is below the inferior turbinate attachment as determined by the nasoendoscopy at screening
11. have a nasal septum perforation
12. have had more than 1 episode of epistaxis with frank bleeding in the month before Visit 1 (Screening)
13. have evidence of significant mucosal injury, ulceration (eg, exposed cartilage) on Visit 1 (Screening) nasal examination/nasoendoscopy
14. have current, ongoing rhinitis medicamentosa (rebound rhinitis)
15. have significant oral structural abnormalities (eg, a cleft palate)
16. have a diagnosis of cystic fibrosis
17. history of eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome) or dyskinetic ciliary syndromes
18. Symptom resolution or last dose of antibiotics for purulent nasal infection, acute sinusitis, or upper respiratory tract infection, influenza, or SARS-CoV-2 (COVID-19) has not occurred before Visit 1 or was less than 4 weeks before the CT scan. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution.
19. planned sinonasal surgery during the period of the study
20. allergy, hypersensitivity, or contraindication to corticosteroids or steroids
21. has used oral steroids in the past for treatment of CRS and did not experience any relief of symptoms
22. has a steroid eluting sinus stent still in place within 30 days of Visit 1
23. allergy or hypersensitivity to any excipients in study drug
24. exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before Visit 1 (Screening); except as noted in inclusion criteria for subjects with comorbid asthma or COPD
25. have nasal candidiasis
26. history or current diagnosis of any form of glaucoma or ocular hypertension
27. history of intraocular pressure (IOP) elevation on any form of steroid therapy
28. history or current diagnosis of the presence (in either eye) of a cataract unless both natural intraocular lenses have been removed
29. history of immunodeficiency
30. any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
31. have a positive drug screen or a recent (within 1 year of Visit 1 [Screening]) history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
32. have participated in an investigational drug clinical trial within 30 days of Visit 1 (Screening)
33. have received mepolizumab (Nucala®), reslizumab (Cinquair®), dupilumab (Dupixent®), omalizumab (Xolair®), or benralizumab (Fasenra™) within 6 months of Visit 1 (Screening)
34. is using strong cytochrome P450 3A4 (CYP3A4) inhibitor (eg, ritonavir, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, saquinavir, ketoconazole, telithromycin, conivaptan, lopinavir, voriconazole, cobicistat)
35. is an employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, or is a family member of the employee or the investigator
36. Patients who report unexplained worsening of vision within the past 3 months (e.g. difficulty reading or seeing traffic signs from a distance.). A diagnosis of presbyopia established by an eye doctor is not exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carothers, Study Director — Optinose US Inc.; John Messina, Study Chair — Optinose US Inc.
Locations (92):
- United States (46):
  - AZ Allergy & Immunology Research, Gilbert, Arizona
  - Kern Research, Bakersfield, California
  - Sacramento Ear, Nose & Throat Surgical and Medical Group Inc, Folsom, California
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Jonathan Corren, MD, Clinical Research Division, Los Angeles, California
  - Sacramento Ear, Nose & Throat, Roseville, California
  - UC Davis Medical Center, Sacramento, California
  - Allergy and Asthma Associates of Santa Clara Valley, San Jose, California
  - Breathe Clear Institute, Torrance, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Yale School of Medicine Section of Otolaryngology, New Haven, Connecticut
  - Emory University MOT, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Midwest Allergy Sinus Asthma, Normal, Illinois
  - Advanced ENT and Allergy, New Albany, Indiana
  - Iowa Head & Neck, Des Moines, Iowa
  - Kentuckiana Ear Nose & Throat, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Ear, Nose and Throat Associates at Greater Baltimore Medical Center, Towson, Maryland
  - St. Cloud Ear, Nose & Throat, Saint Cloud, Minnesota
  - University of Missouri, Dept of Otorlaryngology, Columbia, Missouri
  - Asthma, Allergy, and Immunology Associates, PC, Lincoln, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - ENT and Allergy Associates, New Hyde Park, New York
  - Mount Sinai Downtown Union Square, New York, New York
  - Madison ENT and Facial Plastic Surgery, New York, New York
  - Allergy Asthma & Immunology Relief of Charlotte, Charlotte, North Carolina
  - Allergy Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Research Center, Portland, Oregon
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - Hospital at the University of PA, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - National Allergy and Asthma Research, North Charleston, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - University of TX Health Science Ctr at Houston, Houston, Texas
  - STAAMP Research, LLC, San Antonio, Texas
  - Intermountain Ear, Nose & Throat, Salt Lake City, Utah
  - Chrysallis Clinical Research, St. George, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
  - Spokane ENT, Spokane Valley, Washington
- Bulgaria (6):
  - UMHAT - Kaspela EOOD, Plovdiv
  - MC Iskar, Sofia
  - Multiprofile Hospital for Active Treatment Serdika, Sofia
  - MC Pirogov, Sofia
  - The Military Medical Academy (MHAT), Sofia
  - Мinistry of Interior - Medical Institute, Sofia
- Canada (3):
  - University of British Columbia and Providence Health Care, Vancouver, British Columbia
  - St. Joseph's Healthcare London, London, Ontario
  - CHU de Quebec, pavillon Hopital Saint- Sacrement, Québec
- Georgia (5):
  - Ltd Acad. Fridon Todua Medical Center, Tbilisi
  - Ltd Israel-Georgian Medical Research Clinic - Helsicore, Tbilisi
  - JSC Curatio, Tbilisi
  - Ltd Aversi Clinic, Tbilisi
  - Ltd Simon Khechinashvili University Hospital, Tbilisi
- Poland (15):
  - Jarosław Ślifirski Indywidualna Praktyka Lekarska, Kęty, Lesser Poland Voivodeship
  - Centrum Medyczne Biotamed, Wieliczka, Lesser Poland Voivodeship
  - Medicus Sp z o.o., Wroclaw, Lower Silesian Voivodeship
  - Mini Clinic Paweł Białogłowski, Łańcut, Podkarpackie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - NZOZ Centrum Medyczne LiMED, Tarnowskie Góry, Silesian Voivodeship
  - NZOZ Imedica, Poznan, Wielkopolska
  - ReumaClinic, Bialystok
  - Przychodnia "Narutowicza", Inowrocław
  - Centrum Medyczne All Med - Krakow, Krakow
  - Medical Center Woś i Piwowarczyk, Krakow
  - Centrum Alergologii, Lublin
  - Centrum Medyczne Lucyna Andrazej Dymek - Strzelce Opolskie, Strzelce Opolskie
  - NZOZ "Ignis" dr med. Alicja Łobińska, Świdnik
  - NZOZ Przychodnia Medycyny Rodzinnej, Świętochłowice
- Russia (7):
  - I.M. Sechenov First Moscow State Medical University-University Hospital No.1 - Ear, Nose, and Throat Clinic, Moscow, Moskovskaya Obl.
  - Moscow Regional Scientific Research Clinical Institute n.a. M.F. Vladimirsky (MONIKI), Moscow, Moskovskaya Obl.
  - Saint-Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg, Sankt-Peterburg
  - Smolensk, "Uromed", Smolensk, Smolenskaya Obl
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, Yaroslavskaya Obl.
  - Central Clinical Hospital with Polyclinic" Office of Affairs of the President of the Russian Federation, Moscow
  - Saint-Petersburg Institute of Ear, Nose, Throat, and Speech (The RSFSR Ministry of Health), Saint Petersburg
- Sweden (5):
  - ONH Klinikun Skane Universitetssjukhuset (Lund - Oron- Nas- Och Halskliniken), Lund, Skåne County
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Helsingborg Hospital, Helsingborg, Sverige
  - ONH Kliniken Sahlgrenska Universitetsynkhiset, Gothenburg, Vastra Gotaland Lan
  - Sofiahemmet Hospital, Stockholm
- United Kingdom (5):
  - University Hospital of Wales, Cardiff, CF14 4XW
  - Darlington Memorial Hospital, Darlington
  - Lister Hospital, Stevenage
  - Stockport NHS Foundation Trust (Stepping Hill Hospital Base), Stockport
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPN-375 186 μg BID: OPN-375 186 μg BID x 24 Weeks
  OPN-375: OPN-375, Twice Daily (BID)
- OPN-375 372 μg BID: OPN-375 372 μg BID x 24 Weeks
  OPN-375: OPN-375, Twice Daily (BID)
- Placebo: Matching Placebo BID x 24 Weeks
  OPN-375: OPN-375, Twice Daily (BID)
Period: Overall Study
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Started | 111 | 109 | 112
Completed | 102 | 101 | 96
Not Completed | 9 | 8 | 16
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Lack of Efficacy | 4 | 2 | 9
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Reason not provided | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo | Total
Number analyzed (Participants) | 111 | 109 | 112 | 332
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 93 | 89 | 277
  >=65 years | 16 | 16 | 23 | 55
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 48.4 (13.85) | 49.6 (13.49) | 49.2 (15.26) | 49.1 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 51 | 141
  Male | 64 | 66 | 61 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 9 | 8 | 18
  Not Hispanic or Latino | 110 | 100 | 104 | 314
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 5 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 4 | 6 | 20
  White | 99 | 99 | 101 | 299
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 7 | 7 | 16
  Sweden | 2 | 4 | 2 | 8
  United States | 62 | 64 | 57 | 183
  Poland | 33 | 25 | 32 | 90
  United Kingdom | 0 | 1 | 1 | 2
  Georgia | 2 | 0 | 0 | 2
  Bulgaria | 2 | 3 | 2 | 7
  Russia | 8 | 5 | 11 | 24
Intranasal corticosteroid treatment for chronic sinusitis within the last 10 years [Number; unit: participants]
  Mometason Furoate | 44 | 51 | 48 | 143
  Fluticasone proprionate | 62 | 66 | 67 | 195
  Fluticasone Furoate | 12 | 14 | 20 | 46
  Budesonide | 18 | 22 | 18 | 58
  Ciclesonide | 1 | 1 | 2 | 4
  Beclomethasone | 2 | 7 | 9 | 18
  Triamcinolone | 14 | 11 | 16 | 41
  Flunisolide | 0 | 0 | 1 | 1
  Fluticasone and azelastine | 15 | 14 | 17 | 46
  Other | 6 | 3 | 4 | 13
  Any Treatment | 100 | 100 | 104 | 304
Prior Sinusitis Surgery [Number; unit: participants]
  Any surgery | 58 | 53 | 58 | 169
  Endoscopic sinus surgery | 52 | 47 | 48 | 147
  Balloon sinuplasty | 5 | 4 | 5 | 14
  Polypectomy alone | 14 | 12 | 21 | 47
  Other surgery | 5 | 2 | 3 | 10
  Sinus stent | 2 | 2 | 8 | 12
  Propel mometasone furoate implant | 2 | 2 | 8 | 12
  Sinuva mometasone furoate sinus implant : Yes | 1 | 0 | 0 | 1
Other Chronic Sinusitis Treatment History [Count of Participants; unit: Participants] — History of treatment for Chronic Sinusitis other than corticosteroids and surgery.
  Participants
    Systemic antibiotic in last 5 years: Yes | 44 | 48 | 42 | 134
    Systemic antibiotic in last 5 years: No | 67 | 61 | 70 | 198
    Saline lavage: Yes | 36 | 50 | 39 | 125
    Saline lavage: No | 75 | 59 | 73 | 207
Sinus imaging in last year [Count of Participants; unit: Participants]
  CT scans: 0 | 64 | 59 | 54 | 177
  CT scans: 1 | 40 | 42 | 50 | 132
  CT scans: 2 | 6 | 8 | 8 | 22
  CT scans: 3 | 1 | 0 | 0 | 1
  MRI scans: 0 | 107 | 106 | 105 | 318
  MRI scans: 1 | 4 | 3 | 7 | 14
  MRI scans: 2 | 0 | 0 | 0 | 0
  MRI scans: 3 | 0 | 0 | 0 | 0
Smoking History [Number; unit: participants]
  Current cigarette smoker | 5 | 3 | 6 | 14
  Current smoker (other forms of tobacco) | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptoms as Measured by a Composite Score for Each Symptom of Nasal Congestion, Facial Pain or Pressure Sensation, and Nasal Discharge (Anterior and/or Posterior) at the End of Week 4
Description: Change from baseline to the end of Week 4 in average total instantaneous AM scores (evaluation of symptom severity immediately preceding the time of scoring) for each symptom: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation. Baseline scores are the averaged total instantaneous AM scores over the last 7 days of the single blind run in period, and the end of Week 4, scores are averaged over the 7 days from the subject diary. Range of scores for each nasal symptom is 0= none, 1 = mild, 2 = moderate, 3 = severe. Composite score is a sum of the 3 symptom scores and will range from 0 to 9.
Time Frame: 4 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 108 | 106 | 108
score on a scale | -1.58 (0.161) | -1.60 (0.163) | -0.62 (0.161)

2. Primary Outcome: Change From Baseline to Week 24/Early Termination (ET) in the Average Percent of the Volume Opacified in the Ethmoid and Maxillary Sinuses
Description: Change from baseline to Week 24/ET in the average percent of ethmoid and maxillary sinus volume opacified as measured by CT. Percent volume opacified can range from 0% to 100%. Outcome measure is the percentage change from percent opacification at baseline to percent opacification at Week 24; therefore, change in opacification volume can range from -100% to 100%. For example, if Baseline opacification was 68.22% and Week 24 opacification was 66.11%, then the change would be reported as -2.11%.
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Percentage of volume opacified
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 101 | 99
Percentage of volume opacified | -5.58 (1.436) | -6.20 (1.412) | -1.60 (1.421)

3. Secondary Outcome: Change From Baseline to Defined Timepoint - Subject Symptoms and Functioning as Measured by the Sinonasal Outcome Test - 22-item (SNOT-22) Total Score and Sub Domains
Description: The SNOT-22 is a subject-completed questionnaire that consists of 22 symptoms and social/emotional consequences of their nasal disorder across several domains including: rhinologic, ear/facial pain, psychological dysfunction, and sleep dysfunction. Total scores range from 0-110. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem,3=moderate problem, 4=severe problem, 5=problem as bad as it can be.
Time Frame: Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 96 | 93
score on a scale | -18.05 (1.687) | -22.77 (1.709) | -10.16 (1.723)

4. Secondary Outcome: Change From Baseline in Symptoms as Measured by a Composite Score for Each Symptom of Nasal Congestion, Facial Pain or Pressure Sensation, and Nasal Discharge (Anterior and/or Posterior)
Description: Change from baseline in average total instantaneous AM scores (evaluation of symptom severity immediately preceding the time of scoring) for each symptom: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation. Baseline scores are the averaged total instantaneous AM scores over the last 7 days of the single blind run in period, and the end of Week 4, scores are averaged over the 7 days from the subject diary. Range of scores for each nasal symptom is 0= none, 1 = mild, 2 = moderate, 3 = severe. Composite score is a sum of the 3 symptom scores and will range from 0 to 9.
Time Frame: Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 100 | 99 | 96
score on a scale | -1.89 (0.204) | -2.18 (0.208) | -1.35 (0.208)

5. Secondary Outcome: Change From Baseline in Nasal Congestion Measured by AM and PM Diary Symptom Scores
Description: Subjects will report both instantaneous (evaluation of symptom severity immediately preceding the time of scoring) and reflective (evaluation of symptom severity over the past 12 hours), The Nasal Symptom Scale scores as 0=none, 1=mild-symptoms clearly present but minimal awareness, and easily tolerated, 2= moderate - definite awareness of symptoms that is bothersome but tolerable, 3 = severe - symptoms that are hard to tolerate, cause interference with activities or daily living.
Time Frame: 12 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 100 | 100 | 96
score on a scale
  AM Diary Score: number analyzed (Participants) | 100 | 99 | 96
  AM Diary Score | -0.71 (0.074) | -0.84 (0.076) | -0.45 (0.076)
  PM Diary Score | -0.68 (0.075) | -0.82 (0.076) | -0.41 (0.076)

6. Secondary Outcome: Change in Sense of Smell Scores Measured by AM and PM Diary Symptom Scores
Description: Subjects will report both instantaneous (evaluation of symptom severity immediately preceding the time of scoring) and reflective (evaluation of symptom severity over the past 12 hours) The sense of smell scored as 0= normal, 1=slightly impaired, 2=moderately impaired, 3=absent. The change reported in the results is calculated by subtracting the score reported at Baseline from the score reported at Visit 4 (Week 12).
Time Frame: 12 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 110 | 107 | 110
score on a scale
  AM Diary Score: number analyzed (Participants) | 100 | 99 | 96
  AM Diary Score | -0.60 (0.078) | -0.54 (0.079) | -0.31 (0.079)
  PM Diary Score: number analyzed (Participants) | 100 | 100 | 96
  PM Diary Score | -0.54 (0.078) | -0.56 (0.080) | -0.32 (0.079)

7. Secondary Outcome: Change From Baseline in Nasal Discharge (Anterior and/or Posterior) Measured by AM and PM Diary Symptom Scores
Description: Subjects will report both instantaneous (evaluation of symptom severity immediately preceding the time of scoring) and reflective (evaluation of symptom severity over the past 12 hours). The Nasal Symptom Scale scores as 0=none, 1=mild-symptoms clearly present but minimal awareness, and easily tolerated, 2= moderate - definite awareness of symptoms that is bothersome but tolerable, 3 = severe - symptoms that are hard to tolerate, cause interference with activities or daily living.
Time Frame: 12 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 110 | 107 | 110
score on a scale
  AM Diary Score: number analyzed (Participants) | 100 | 99 | 96
  AM Diary Score | -0.65 (0.075) | -0.74 (0.076) | -0.43 (0.077)
  PM Diary Score: number analyzed (Participants) | 100 | 100 | 96
  PM Diary Score | -0.58 (0.077) | -0.72 (0.078) | -0.37 (0.078)

8. Secondary Outcome: Change in Facial Pain or Pressure Sensation Measured by AM and PM Diary Symptom Scores
Description: Subjects will report both instantaneous (evaluation of symptom severity immediately preceding the time of scoring) and reflective (evaluation of symptom severity over the past 12 hours). The Nasal Symptom Scale scores as 0=none, 1=mild-symptoms clearly present but minimal awareness, and easily tolerated, 2= moderate - definite awareness of symptoms that is bothersome but tolerable, 3 = severe - symptoms that are hard to tolerate, cause interference with activities or daily living.
  The value reported in the results is calculated by subtracting the score reported by the patient at Baseline from the score reported by the patient at Visit 4 (Week 12).
Time Frame: 12 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 110 | 107 | 110
score on a scale
  AM Diary Score: number analyzed (Participants) | 100 | 99 | 96
  AM Diary Score | -0.53 (0.078) | -0.61 (0.079) | -0.48 (0.079)
  PM Diary Score: number analyzed (Participants) | 100 | 100 | 96
  PM Diary Score | -0.52 (0.077) | -0.57 (0.079) | -0.43 (0.078)

9. Secondary Outcome: Change From Baseline to Week 24/Early Termination (ET) in the Average Percent of the Volume Opacified in the Ethmoid and Maxillary Sinuses Among Patient Populations
Description: Change from baseline to Week 24/ET in the average percent of ethmoid and maxillary sinus volume opacified as measured by CT for CRS with Nasal Polyps (NP) and without NP sub-groups and in patients with and without previous sinus surgery. Percent volume opacified can range from 0% to 100%. Outcome measure is percentage change from percent opacification at baseline to percent opacification at Week 24; therefor, change in opacification volume can range from -100% to 100%. For example, if Baseline opacification was 68.22% and Week 24 opacification was 66.11%, then the change would be reported as -2.11%.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of volume opacified
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 101 | 99
percentage of volume opacified
  Nasal Polyps Present: number analyzed (Participants) | 63 | 63 | 62
  Nasal Polyps Present | -6.01 (1.741) | -4.64 (1.744) | 1.29 (1.727)
  Nasal Polyps Absent: number analyzed (Participants) | 35 | 38 | 37
  Nasal Polyps Absent | -3.52 (2.389) | -7.90 (2.287) | -5.50 (2.309)
  Prior Sinus Surgery: number analyzed (Participants) | 45 | 40 | 41
  Prior Sinus Surgery | -7.58 (2.156) | -8.91 (2.235) | -1.65 (2.185)
  No Prior Sinus Surgery: number analyzed (Participants) | 53 | 61 | 58
  No Prior Sinus Surgery | -3.30 (1.913) | -3.82 (1.787) | -0.95 (1.810)

10. Secondary Outcome: Change From Baseline to Week 24/ET in the Lund-Mackay Staging System Total Score
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification), plus a 0-2 score for each of the left and right ostiomeatal complex (OMC). The total LM score for a CT scan ranges from 0-24.
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale | -0.40 (0.269) | -0.46 (0.267) | 0.10 (0.266)

11. Secondary Outcome: Change From Baseline to Week24/ET in the Lund-Mackay Staging System Total Scores for Ethmoids and Maxillary Sinuses Combined
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification), plus a 0-2 score for the ostiomeatal complex (OMC).
  The values reported for this outcome are the change in total opacification of the left and right maxillary and ethmoid sinuses (Visit 6 [Wk 24] score minus Baseline score). Each visit score can range from a total of 0-12 (sum of 0-2 score assigned for each of left and right maxillary, left and right anterior ethmoid, and left and right posterior ethmoid).
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale | 0.12 (0.148) | 0.04 (0.149) | 0.37 (0.148)

12. Secondary Outcome: Change From Baseline to Week24/ET in the Lund-Mackay Staging System Total Scores for Sinus Pairs
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification), plus a 0-2 score for the ostiomeatal complex (OMC).
  Each sinus pair (left and right side) listed below can achieve a total score of 0-4 (sum of 0-2 for each side). The values reported below are calculated by subtracting the total score at Baseline from the total score at Visit 6 (Wk 24).
Time Frame: Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale
  Ethmoid Sinus Anterior | 0.06 (0.064) | -0.01 (0.063) | 0.07 (0.064)
  Ethmoid Sinus Posterior | 0.00 (0.066) | -0.04 (0.067) | 0.15 (0.068)
  Maxillary Sinus | 0.04 (0.049) | 0.09 (0.051) | 0.12 (0.052)
  Frontal Sinus | 0.08 (0.072) | 0.01 (0.071) | 0.01 (0.070)
  Sphenoid Sinus | 0.04 (0.067) | -0.03 (0.068) | 0.08 (0.069)
  Ostiomeatal Complex | -0.66 (0.129) | -0.47 (0.129) | -0.31 (0.129)

13. Secondary Outcome: Change From Baseline to Week 24/ET in Average Percent of Sinus Volume Occupied by Disease in the Worst Maxillary Sinus as Measured by CT Scan Assessment
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Percent opacified volume
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 101 | 99
Percent opacified volume | -14.70 (2.23) | -12.62 (2.3) | -7.61 (2.29)

14. Secondary Outcome: Change From Baseline to Week 24/ET in Average Percent of Sinus Volume Occupied by Disease in the Worst Ethmoid Sinus as Measured by CT Scan Assessment
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Percent opacified volume
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 101 | 99
Percent opacified volume | -7.31 (1.43) | -7.43 (1.44) | -3.76 (1.44)

15. Secondary Outcome: Change From Baseline to Week 24/ET in Average Percent of Sinus Volume Occupied by Disease in the Worst Sinus Between the Maxillary and Ethmoid Sinuses as Measured by CT Scan Assessment Among Patient Populations
Description: Percent of sinus volume occupied by disease in the worst sinus between maxillary and ethmoid sinuses for the total population, chronic rhinosinusitis with nasal polyps (CRSwNP) subgroup, chronic rhinosinusitis without nasal polyps (CRSsNP) subgroup, patients with previous sinus surgery subgroup, and without previous surgery subgroup.
Time Frame: 24 Weeks
Population: Data is provided for the total population and 4 subgroups. The population of the subgroups will not equal the total population, as they are only a portion of subjects from the total.
Measure: Least Squares Mean (Standard Error); unit: Percent opacified volume
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 98 | 101 | 99
Percent opacified volume
  Full Population | -11.27 (1.81) | -10.39 (1.83) | -6.51 (1.82)
  CRSwNP SubGroup: number analyzed (Participants) | 63 | 63 | 62
  CRSwNP SubGroup | -6.54 (1.77) | -6.72 (1.81) | -3.23 (1.79)
  CRSsNP SubGroup: number analyzed (Participants) | 35 | 38 | 37
  CRSsNP SubGroup | -7.88 (2.37) | -7.89 (2.37) | -3.88 (2.34)
  Subjects with Prior Sinus Surgery: number analyzed (Participants) | 45 | 40 | 41
  Subjects with Prior Sinus Surgery | -11.29 (2.67) | -12.44 (2.89) | -3.24 (2.85)
  Subjects without Prior Sinus Surgery: number analyzed (Participants) | 53 | 61 | 58
  Subjects without Prior Sinus Surgery | -11.00 (2.46) | -8.83 (2.30) | -8.39 (2.33)

16. Secondary Outcome: Change From Baseline to Week 24/ET in the Zeinrich Modification of Lund-Mackay Staging System Total Score
Description: Zeinrich Modification of the Lund-Mackay Staging System:
  Zeinrich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100% for each sinus. Total score ranges from 0 to 50.
Time Frame: Baseline, Week 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale | -0.98 (0.65) | -1.95 (0.64) | -0.03 (0.65)

17. Secondary Outcome: Change From Baseline to Week 24/ET in the Zeinrich Modification of Lund-Mackay Staging System for Ethmoids and Maxillary Sinuses Combined
Description: Zeinrich Modification of the Lund-Mackay Staging System:
  Zeinrich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100% The total score for the combined ethmoids and maxillary sinuses can range from 0-30 (0-5 for each left and right of the anterior ethmoid, posterior ethmoid, and maxillary sinuses). The outcome values presented in the results are determined by subtracting the total score at Baseline from the total score at Week 24.
Time Frame: Baseline, Week 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale | -1.21 (0.43) | -1.44 (0.43) | -0.19 (0.42)

18. Secondary Outcome: Change From Baseline to Week 24/ET in the Zeinrich Modification of Lund-Mackay Staging System for the Sinus Pairs
Description: Zeinrich Modification of the Lund-Mackay Staging System:
  Zeinrich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100% Each sinus pair (left and right side) listed below can achieve a total score of 0-10 (sum of score on each side). The values reported for this outcome calculated by subtracting the score at Baseline from the score at Visit 6 (Wk 24).
Time Frame: Baseline, Week 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale
  Anterior Ethmoid Sinus Pair | -0.39 (0.17) | -0.53 (0.17) | -0.19 (0.17)
  Posterior Ethmoid Sinus Pair | -0.33 (0.18) | -0.55 (0.18) | 0.03 (0.18)
  Maxillary Sinus Pair | -0.53 (0.18) | -0.39 (0.17) | -0.08 (0.17)
  Frontal Sinus Pair | 0.12 (0.20) | -0.16 (0.20) | 0.05 (0.20)
  Sphenoid Sinus Pair | 0.15 (0.20) | -0.16 (0.19) | 0.20 (0.19)

19. Secondary Outcome: Change From Baseline to Week 24/ET in the Zeinrich Modification of Lund-Mackay Staging System for the Worst Sinus Between Maxillary and Ethmoid Sinuses Among Patient Populations
Description: Zeinrich Modification of the Lund-Mackay Staging System:
  Zeinrich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100%
Time Frame: Baseline, Week 24
Population: Data provided for full population and CRSwNP, CRSsNP, subjects with prior sinus surgery, and subjects without prior sinus surgery subgroups. Number of participants analyzed in the subgroups will be less than the total overall, as these are only portions of the total population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 101 | 99
score on a scale
  Total Population | -0.59 (0.11) | -0.60 (0.11) | -0.45 (0.11)
  CRSwNP: number analyzed (Participants) | 63 | 63 | 62
  CRSwNP | -0.49 (0.13) | -0.57 (0.14) | -0.30 (0.14)
  CRSsNP: number analyzed (Participants) | 36 | 38 | 37
  CRSsNP | -0.70 (0.18) | -0.61 (0.18) | -0.64 (0.18)
  Subjects with Prior Sinus Surgery: number analyzed (Participants) | 45 | 40 | 41
  Subjects with Prior Sinus Surgery | -0.48 (0.16) | -0.78 (0.17) | -0.33 (0.17)
  Subjects without Prior Sinus Surgery: number analyzed (Participants) | 54 | 61 | 58
  Subjects without Prior Sinus Surgery | -0.70 (0.15) | -0.51 (0.14) | -0.54 (0.14)

20. Secondary Outcome: Time Comparison to First Acute Exacerbation of Chronic Sinusitis
Description: Comparing the distribution of time to first acute exacerbation of chronic sinusitis, defined as a worsening of symptoms that requires escalation of treatment
Time Frame: 24 Weeks
Population: Number of patients experiencing exacerbation within each treatment group.
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 17 | 7 | 21
Weeks | 23.44 (0.55) | 17.19 (0.25) | 19.73 (0.69)

21. Secondary Outcome: Percentage of Subjects Requiring Rescue Medication After Week 4
Description: Recording of each dose of approved rescue medication after the Week 4 visit through Week 12
Time Frame: 8 Weeks
Population: We were unable to complete this analysis due to a misunderstanding on the part of the subjects in the definition of "rescue medication". It was confirmed across most countries and sites that subjects indicated use of rescue medication mistakenly, thinking they were being asked to report whether they took the study medication. This data could not be fully reconciled and, therefore, no analysis was completed.
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Change in Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a validated, self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate 7 "component" scores (each ranging between 0 and 3): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these 7 components yields 1 global score ranging between 0 and 21. Higher values represent a worse outcome.
Time Frame: 12 Weeks, 24 Weeks
Population: Full analysis set. Population sizes differ based on number of patients that completed the assessment at each timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 99 | 98 | 96
score on a scale
  Week 12: number analyzed (Participants) | 97 | 98 | 96
  Week 12 | -0.66 (0.291) | -1.48 (0.291) | -0.91 (0.294)
  Week 24: number analyzed (Participants) | 99 | 97 | 92
  Week 24 | -1.12 (0.292) | -1.77 (0.294) | -1.09 (0.301)

23. Secondary Outcome: Change in Overall Health From Baseline to Week 4 and Week 24/ET as Measured by the Percent of Subjects Improved as Indicated by the Patient Global Impression of Change (PGIC)
Description: Global impression of change will be assessed using a subject-completed PGIC scale range: 1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse
Time Frame: Week 4, Week 24
Population: Population size at each timepoint differs based on the number of patients that completed the assessment at the timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 109 | 103 | 104
Participants
  Week 4 | 84 | 77 | 57
  Week 24: number analyzed (Participants) | 99 | 98 | 94
  Week 24 | 78 | 80 | 56

24. Secondary Outcome: Severity of Depression at Week 24 as Measured by the Quick Inventory of Depression Symptomatology (QIDS)
Description: The 16-item QIDS (Rush et al. 2003) is designed to assess the severity of depressive symptoms. The QIDS is available in a self-rated version and assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 5th edition to diagnose a major depressive episode. The 7-day period prior to assessment is the usual time frame for assessing symptom severity. Scores range from 0 to 27, where higher scores indicate a worse outcome.
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 102 | 101 | 100
score on a scale | -0.24 (0.31) | -0.80 (0.31) | -0.62 (0.31)

25. Secondary Outcome: Change in the 36-Item Short Form Health Survey Version 2 (SF-36v2) Mental Composite Score (MCS)
Description: Change from baseline to Week 24/ET on the MCS of the 36-Item Short Form Health Survey version 2 (SF-36v2). The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire. The scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: 24 Weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 101 | 101 | 101
score on a scale | -0.1 (0.810) | 1.65 (0.820) | 1.41 (0.834)

26. Secondary Outcome: Change in the SF-36v2 Physical Composite Score (PCS)
Description: Change from baseline to Week 24/ET on the PCS of the 36-Item Short Form Health Survey version 2 (SF-36v2). The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire. The scale range is from 0-100. A lower score means more disability and a higher score means less disability.
Time Frame: 24 Weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 101 | 101 | 101
score on a scale | 2.37 (0.647) | 3.64 (0.652) | 1.58 (0.663)

27. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Short-Form 36 Health Survey, Version 2 (SF-36v2)
Description: The SF-36v2 is a multipurpose, 36-item subject-completed validated questionnaire that measures 8 domains of health: physical functioning, role limitations due to physical health (RP), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The SF-36v2 survey with a 4-week recall will be used. It yields scale scores for each of these 8 health domains , each of which is scored from 0 to 100. Higher scores indicate with a better health status, with 100 representing the highest level of functioning possible.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 102 | 101 | 101
score on a scale
  Physical Functioning Score | 1.07 (1.039) | 1.43 (1.055) | 0.04 (1.067)
  Role Physical Score | 0.92 (1.057) | 2.64 (1.074) | 0.16 (1.082)
  Bodily Pain Score | 0.94 (1.172) | 4.10 (1.185) | 1.8 (1.201)
  General Health Score | 0.55 (1.091) | 2.38 (1.119) | -1.18 (1.21)
  Vitality Score | 1.13 (1.142) | 3.35 (1.156) | 1.81 (1.168)
  Social Functioning Score | 0.22 (1.153) | 2.05 (1.173) | 1.89 (1.181)
  Role Emotional Score | -1.11 (1.147) | 1.2 (1.169) | -0.32 (1.178)
  Mental Health Score | -0.92 (1.169) | 0.75 (1.188) | -0.69 (1.194)

28. Secondary Outcome: Change in Depressive Symptoms From Baseline to Week 24/ET as Measured by Change in the Severity of Depression as Measured by the Quick Inventory of Depression Symptomatology (QIDS)
Description: The 16-item QIDS (Rush et al. 2003) is designed to assess the severity of depressive symptoms. The QIDS is available in a self-rated version and assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 5th edition to diagnose a major depressive episode. The 7-day period prior to assessment is the usual time frame for assessing symptom severity. Scores range from 0 to 27, with higher scores indicating a worse outcome.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 102 | 101 | 100
score on a scale | -0.24 (0.308) | -0.80 (0.312) | -0.62 (0.314)

29. Secondary Outcome: Change in Olfactory Impairment From Baseline to Week 24/ET as Measured by the Smell Identification Test (SIT)™
Description: The SIT is a test comprised of 4 booklets each containing 10 microencapsulated (scratch and sniff) odors. Forced choice response alternatives to identify the odor accompany each test item. Each correct response is assigned a score of 1 and incorrect responses are assigned a score of 0. The total score is calculated by summing the scores of each individual odor for a total possible score ranging from 0-40. The higher the score, the better the individual's sense of smell. The test provides an absolute indication of smell loss (anosmia; mild, moderate or severe hyposmia) as well as an index to detect malingering.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 100 | 100 | 93
score on a scale | 2.47 (0.765) | 2.33 (0.768) | -1.30 (0.793)

30. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Euroqol 5-dimension (EQ-5D) Instrument Visual Analogue Scale (VAS)
Description: The EQ-5D consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The outcome measured for this study was the EQ VAS, which records the subject's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the subject's own judgement. VAS scores range from 0 (worst health you can imagine) to 100 (best health you can imagine).
Time Frame: 24 Weeks
Population: Full Analysis Set. Only VAS Scores analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 101 | 101 | 100
score on a scale | 2.59 (1.783) | 3.97 (1.791) | -0.35 (1.810)

31. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Short-Form 6-Dimension (SF-6D) Instrument
Description: The SF-6D is a single health state index derived from the 11 items from the SF-36v2. SF-6D scores range from 0 (worst health state) to 1 (best health state).
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 101 | 100 | 101
score on a scale | 0 (0.016) | 0.04 (0.017) | 0.01 (0.016)

32. Secondary Outcome: Comparison of Health Economic Measures- Percentage of Subjects Indicating That They Are Willing to Consider Sinus Surgery
Description: Percentage of subjects indicating that they are willing to consider Sinus Surgery
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 104 | 104 | 102
Participants
  Baseline | 63 | 59 | 54
  Week 24 | 52 | 48 | 54

33. Secondary Outcome: Comparison of Health Economic Measures- Percentage of Subjects Who Meet the Minimal Objective Criteria for Surgical Intervention
Description: Percentage of Subjects who meet the minimal objective criteria for surgical intervention
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 100 | 101 | 102
Participants
  Baseline | 42 | 48 | 45
  Week 24 | 30 | 36 | 38

34. Secondary Outcome: Comparison of Health Economic Measures- Percentage of Subjects Approved for Surgery Who no Longer Elect to Undergo a Surgery
Description: Outcome value presented here is the percent of subjects who are approved for surgery but no longer elect to undergo a surgery. The number of participants analyzed indicates the total number of participants for whom this analysis was completed.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 104 | 104 | 102
Participants | 52 | 56 | 48

35. Secondary Outcome: Change in Work Productivity From Baseline to Week 24/ET as Measured by the Health and Work Performance Questionnaire (HPQ).
Description: The Health and Work Performance Questionnaire measures work productivity (absenteeism and presenteeism). - Absenteeism is measured in missed work days over the past four weeks (range 0-20); absenteeism is measured in % productivity at work (0-100%), with higher values indicating improved productivity. Values for this outcome are reported as the change in relative absenteeism (the percentage of productivity at work) from baseline to Week 24.
Time Frame: 24 Weeks
Population: Full analysis set. Population size determined by the number of patients that completed the questionnaire at baseline and Week 24.
Measure: Mean (Standard Error); unit: percentage of productivity
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 81 | 76 | 75
percentage of productivity | 0.98 (2.384) | -4.13 (2.479) | -6.28 (2.505)

36. Other Pre Specified Outcome: Evaluation of Safety by Recording the Severity of Adverse Events (AEs)
Description: Assessment of safety by measuring severity of AEs using scale with 1=mild, 2=moderate, 3=severe
Time Frame: 24 Weeks
Population: Safety Analysis Set - Subjects with at least 1 AE
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
Participants
  Mild | 25 | 23 | 20
  Moderate | 29 | 26 | 33
  Severe | 3 | 3 | 5

37. Other Pre Specified Outcome: Evaluation of Safety-Nasal Examination
Description: Assessed in nasal examination worksheet which includes recording the presence of any epistaxis, septal erosion/perforation, ulceration/erosion of area other than septum.
Time Frame: 24 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 108 | 105 | 103
Participants
  Epistaxis: Present | 3 | 9 | 1
  Epistaxis: Absent | 105 | 96 | 102
  Septal Erosion/Perforation: Present | 3 | 3 | 0
  Septal Erosion/Perforation: Absent | 105 | 102 | 103
  Ulceration/Erosion (non-septum): Present | 0 | 2 | 1
  Ulceration/Erosion (non-septum): Absent | 108 | 103 | 102
  Mucosal Candidiasis: Present | 0 | 0 | 0
  Mucosal Candidiasis: Absent | 108 | 105 | 103

38. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Blood Pressure
Description: Includes systolic and diastolic blood pressure measurements in millimeter of mercury (mmHg)
Time Frame: 24 Weeks
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 109 | 106 | 104
mmHg
  Systolic Blood Pressure (mmHg) | 127.3 (14.15) | 126.7 (14.11) | 127.3 (14.69)
  Diastolic Blood Pressure (mmHg) | 78.0 (8.22) | 78.2 (9.70) | 79.3 (8.62)

39. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Pulse
Description: Measure pulse in beats per minute (bpm)
Time Frame: 24 Weeks
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 109 | 106 | 104
Beats per minute | 73.7 (11.96) | 72.7 (9.5) | 73.1 (9.45)

40. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Weight
Description: Assessment of safety from physical examination-weight measured in kg or lb
Time Frame: 24 Weeks
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 109 | 104 | 104
kg | 82.81 (20.873) | 84.23 (19.232) | 83.84 (21.531)

41. Other Pre Specified Outcome: Evaluation of Safety - Monitoring Concomitant Medication Usage
Description: Assessment for safety from the collection of information for concomitant medications usage
Time Frame: 24 Weeks
Population: Number of subjects receiving concomitant medications. Only top 5 con-meds are detailed below.
Measure: Number; unit: Participants
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
Number analyzed (Participants) | 103 | 100 | 105
Participants
  Amides | 33 | 38 | 30
  Adrenergics in Combination with Corticosteroids or other drugs | 35 | 30 | 27
  Ace Inhibitors, Plain | 5 | 7 | 12
  Allergen Extracts | 6 | 6 | 2
  Alpha-Adrenoreceptor Antagonists | 1 | 6 | 2

ADVERSE EVENTS:
Time Frame: Pretreatment (Screening/Run-in) period to end of treatment (Week 24)
Arm/Group | OPN-375 186 μg BID | OPN-375 372 μg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/109 | 0/112
Serious Adverse Events (participants affected / at risk) | 1/111 | 2/109 | 3/112
Other Adverse Events (participants affected / at risk) | 37/111 | 37/109 | 14/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPN-375 186 μg BID (N=111) | OPN-375 372 μg BID (N=109) | Placebo (N=112)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPN-375 186 μg BID (N=111) | OPN-375 372 μg BID (N=109) | Placebo (N=112)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 13 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Headache (Nervous system disorders) | 2 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 0
Cataract nuclear (Eye disorders) | 5 | 4 | 0
Cataract cortical (Eye disorders) | 6 | 2 | 1
Nasopharyngitis (Infections and infestations) | 6 | 3 | 3
Acute sinusitis (Infections and infestations) | 5 | 2 | 4
Influenza (Infections and infestations) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03781804/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03781804/SAP_001.pdf